CLINICAL TRIAL: NCT03400423
Title: The Acute Effects of Moderate Intensity Exercise and Caffeine Ingestion on Cognition in Non-Caffeine Consumers and Caffeine Consumers
Brief Title: The Acute Effects of Caffeine on Exercise and Cognition
Acronym: AEC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Dr. Harry Prapavessis, Professor, Western University, Canada
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Acute Exercise and Caffeine
Record Dates: First submitted 2018-01-09; First posted 2018-01-17 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2018-01

CONDITIONS: Adult Population
Keywords: Caffeine; Caffeine Withdrawal; Acute Aerobic Exercise; Cognition; Working Memory
MeSH Terms: interventions — Caffeine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Non-caffeine exercise (Experimental): Exercise cognition score
  Interventions: Behavioral: Moderate Intensity Exercise
- Non-caffeine cognition (Active Comparator): Caffeine cognition score
  Interventions: Drug: Caffeine
- Caffeine consumption exercise (Experimental): Exercise cognition score
  Interventions: Behavioral: Moderate Intensity Exercise
- Caffeine consumption cognition (Active Comparator): Caffeine cognition score
  Interventions: Drug: Caffeine
- Deprived Caffeine consumers exercise (Experimental): Exercise cognition score
  Interventions: Behavioral: Moderate Intensity Exercise
- Deprived caffeine consumers cognition (Active Comparator): Caffeine administration cognition score
  Interventions: Drug: Caffeine

INTERVENTIONS:
Drug: Caffeine — Oral administration of 1.2mg/kg of powdered caffeine with water.
  Arms: Caffeine consumption cognition; Deprived caffeine consumers cognition; Non-caffeine cognition
Behavioral: Moderate Intensity Exercise — Moderate intensity exercise conducted on a treadmill. Moderate intensity exercise defined as (220-age)*0.6.
  Arms: Caffeine consumption exercise; Deprived Caffeine consumers exercise; Non-caffeine exercise

SUMMARY:
The effects of moderate intensity aerobic exercise and caffeine ingestion on cognition (more specifically working memory) in non-caffeine drinker and caffeine drinkers will be examined. The non-caffeine drinkers will be recruited for two visits, whereas, the caffeine drinkers will be recruited for three visits. The study involves a baseline assessment of cognition and examines the effects of exercise and caffeine. Finally the caffeine group will consist of a baseline and intervention assessment when deprived of caffeine (overnight abstinence). The exercise intervention is to complete 20-minutes of moderate intensity exercise (brisk walk) while the caffeine condition is to consume 1.2 mg/kg of caffeine. Immediately following both intervention the n-back assessment will be conducted.

DETAILED DESCRIPTION:
Phase 1 will assess non-caffeine consumers

Phase 1 will utilize a within subjects counter-balanced design. Previous to arrival for phase 1, participants will be asked to abstain from alcohol and drugs for at least 18 hours previous. Participants will be urged to arrive at the same time for each visit. Upon arrival to the Exercise and Health Psychology lab (located in room 408 of the Arthur and Sonia Labatt Health Science Building at Western University) participants will be given the letter of information, and asked to sign the informed consent form. After consent, participants will also be asked to complete a demographic survey, PAR-Q readiness for exercise, Godin Leisure-Time Exercise Questionnaire, caffeine consumption questionnaire-R (CCQ-R) and a caffeine withdrawal questionnaire (CWSQ). Vitals (heart rate and blood pressure) will be assessed following the completion of the questionnaires as well as post intervention in the seated position. Prior to evaluation on the N-back task (cognitive memory task described below) a practice stage with be conducted until the participant can consistently score 75% or higher on three consecutive trials to eliminate a learning effect. After establishing test familiarity, a baseline cognition score will be conducted through the n-back assessment. The subject will then be given a 5-minute break (i.e., to use the lavatory). Following the break, the participants will be randomized into either moderate intensity exercise or caffeine ingestion group. The interventions are as follows; Moderate Intensity Exercise will consist of a 20-minute bout of moderate intensity aerobic exercise. Exercise will consist of a 2-minute warm-up, followed by 15 minutes of walking at a rate, which will allow you to reach 2/3 of your max heart rate ((220-age)x0.6) followed by a 3-minute cool down on a treadmill (together equaling 20 minutes). HR will be monitored through heart rate monitors worn by the participants. The caffeine ingestion group will ingest 1.2 mg/kg of caffeine orally in powder form with water to drink, after ingestion of caffeine participants will wait 20 minutes to ensure peak plasma levels. The participants both the exercise group and the caffeine ingestion group will be asked to refrain from conversation. The post intervention assessment will begin within two minutes of the completion of either intervention. The second visit of phase I will take place the following day at the same time (if possible). During the second visit the participant's will complete the pre caffeine or pre exercise questionnaire, the CWSQ and vitals will be monitored pre and post intervention. The participants will participate in the intervention that they have not received on the first visit (for example, if the participant received caffeine ingestion on the first visit the participant will receive moderate intensity aerobic exercise on the second visit). Within two minutes of completion the post treatment N-back task assessment will begin.

Phases 2 and 3 will assess caffeine consumers (phase 3 in an acutely deprived state)

Phase 2 will utilize a within subjects counter-balanced design. Previous to arrival for phase 2 participants will be asked to keep consumption of caffeine to a regular dose (morning coffee) on the day of testing, abstain from alcohol and drugs for at least 18 hours prior to testing. Participants will be urged to arrive at the same time for each visit. Upon arrival to the Exercise and Health Psychology lab (located in room 408 of the Arthur and Sonia Labatt Health Science Building at Western University) participants will be given the letter of information, and asked to sign the informed consent form. Participants will also be asked to complete a demographic survey, PAR-Q readiness for exercise, Godin Leisure-Time Exercise Questionnaire, CCQ-R, and the CWSQ. Vitals (heart rate and blood pressure) will be assessed following the completion of the questionnaires as well as post intervention in the seated position. Prior to evaluation on the N-back task (cognitive memory task described below) a practice stage with be conducted until the participant can consistently score 75% or higher on three consecutive trials to eliminate a learning effect. After establishing familiarity, a baseline cognition score will be conducted through the n-back assessment. The subject will then be given a 5 minute break (i.e., to use the lavatory). Following the break the participants will be randomized into either the moderate intensity exercise or caffeine ingestion group. The interventions are as followed; Moderate Intensity Exercise will consist of a 20-minute bout of moderate intensity aerobic exercise. Exercise will consist of a 2-minute warm-up, followed by 15 minutes of walking at a rate, which will allow you to reach 2/3 of your max heart rate (moderate intensity exercise= (220-age) x 0.6), and then a 3-minute cool down on a treadmill (together equaling 20 minutes). HR will be monitored through heart rate monitors worn by the participants. The caffeine ingestion group will ingest 1.2 mg/kg of caffeine in powder form with water to drink, after ingestion of caffeine participants will wait 20 minutes to ensure peak plasma levels.The participants in both the, exercise group and caffeine ingestion group will be asked to refrain from conversation. The post intervention assessment will begin within two minutes of the completion of either intervention. The second visit of phase I will take place the following day at the same time (if possible). During the second visit the participant's will complete the pre caffeine or pre exercise questionnaire, the CWSQ and vitals will be monitored pre and post intervention. The participants will participate in the intervention that they have not received on the first visit (for example, if the participant received caffeine ingestion on the first visit the participant will receive moderate intensity aerobic exercise on the second visit). Within two minutes of completion the post treatment N-back task assessment will begin.

Prior to arrival for phase 3, participants will be asked to refrain from caffeine for at least 12 hours, and abstain from alcohol and drugs for at least 18 hours prior to testing. Phase 3 will utilize the same participants as phase 2, but they will be examined in a caffeine-deprived state (12 hours) for baseline N-back scores the CWSQ will also be administered. Participants will then be randomized into either the caffeine ingestion group or exercise treatment group where post intervention N-back scores will be obtained. Participants will be asked to complete the same pre-intervention questionnaires as the previous phase. Vitals (heart rate and blood pressure) will be assessed pre and post intervention. Caffeine abstinence will be validated through self-report with the use of deception (participants being told that their saliva sample is being tested for the presence of caffeine).

N-back task explanation: Three tasks will be administered to subjects for each treatment condition (after caffeine administration and after exercise). The 1-back, 2-back, and 3-back cognitive tests will assess working memory by measuring both the percentage of correct responses, as well as reaction time. In these 5 minute tasks, a letter will appear on a computer screen for an interval of 500ms, followed by a 2000ms blank screen interstimulus (totaling 120 letters/5 minutes). Participants will be instructed to click the left button of a computer mouse as soon as a target appears, and to keep in mind both the speed and accuracy components of the task. In the 1-back condition, the target is defined as a letter flashing that is the same as the one preceding it. For example, "x, interstimulus, x" would be the target. In the 2-back condition, the target is defined as a letter appearing that is the same as what preceded it 2 letters before. For example, "a, interstimulus, b, interstimulus, a", would be the target. In the 3-back condition, the target is defined as a letter appearing that is the same as what preceded it 3 letters before. For example, "a, interstimulus, b, interstimulus, c, interstimulus, a", would be the target. All tasks call into action the participant's working memory abilities, as a measure of cognition.

ELIGIBILITY:
Inclusion Criteria:

* Are over the age of 18 years (male or female)
* Do not consume more than 100 mg of caffeine a week
* Do not have any cognitive problems
* Are not pregnant
* Do not have a medical condition that prevents you to exercise
* Do not have an orthopaedic limitation
* Have access to a telephone or an email account for communication
* Can read and write in English You are being invited to take part in phase 2 and 3 of this research study because
* Are over the age of 18 years old
* Are consuming at least 150 mg of caffeine a day
* Do not have any cognitive problems
* Are not pregnant
* Do not have a medical condition that prevents you to exercise
* Do not have an orthopaedic limitation
* Have access to a telephone or an email account for communication
* Can read and write in English

Exclusion Criteria:

Potential subjects will be excluded if they are pregnant. Additionally, participants taking prescription medication for depression or anxiety, and participants that cannot give informed consent will be excluded.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
3-back on the N-back task | Approximately 5 minutes
  Participants will be instructed to click the left button of a computer mouse as soon as a target appears, and to keep in mind both the speed and accuracy components of the task. In the 1-back condition, the target is defined as a letter flashing that is the same as the one preceding it. For example, "x, interstimulus, x" would be the target. In the 2-back condition, the target is defined as a letter appearing that is the same as what preceded it 2 letters before. For example, "a, interstimulus, b, interstimulus, a", would be the target. In the 3-back condition, the target is defined as a letter appearing that is the same as what preceded it 3 letters before. For example, "a, interstimulus, b, interstimulus, c, interstimulus, a", would be the target. All tasks call into action the participant's working memory abilities, as a measure of cognition.

SECONDARY OUTCOMES:
0,1, and 2 back on the N-back task | Approximately 15 minutes
  Participants will be instructed to click the left button of a computer mouse as soon as a target appears, and to keep in mind both the speed and accuracy components of the task. In the 1-back condition, the target is defined as a letter flashing that is the same as the one preceding it. For example, "x, interstimulus, x" would be the target. In the 2-back condition, the target is defined as a letter appearing that is the same as what preceded it 2 letters before. For example, "a, interstimulus, b, interstimulus, a", would be the target. In the 3-back condition, the target is defined as a letter appearing that is the same as what preceded it 3 letters before. For example, "a, interstimulus, b, interstimulus, c, interstimulus, a", would be the target. All tasks call into action the participant's working memory abilities, as a measure of cognition.

CONTACTS AND LOCATIONS:
Locations (1):
- Western University, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
We do not plan to share IPD.